CLINICAL TRIAL: NCT07237152
Title: Risk Factors for Chronic Limb Pain in Major Trauma Patients With Limb Injury
Brief Title: Chronic Pain Predictors in Major Trauma
Acronym: COPE: MT
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 25034
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain; Limb Fracture
Keywords: chronic pain; limb fracture; risk factors; prediction model
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about who is at risk of developing chronic pain in a major trauma population with at least one limb fracture.

The main question it aims to answer is: which risk factors predict which patients will experience chronic pain following traumatic limb injury.

Participants will answer a baseline questionnaire and two outcome questionnaires about their pain at 3 and 6 months after their injury.

ELIGIBILITY:
Inclusion Criteria:

Aged ≥ 16 Polytrauma patient (multiple injuries affecting multiple body regions or organ systems) Admitted to a UK Major Trauma Centre Minimum of 1 radiologically confirmed traumatic limb fracture Have capacity to provide informed consent to participate in the study Have sufficient proficiency in English to provide the required data or be willing to use an approved interpreting service for data collection Recruited within 4 weeks of injury

Exclusion Criteria:

No traumatic limb fracture Patients with a primary or treatment amputation in relation to their limb injury Pathological limb fractures Prisoners No fixed abode

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult major trauma patients with a minimum of one limb fracture treated at the East Midlands Major Trauma Centre based at Nottingham University Hospitals NHS Trust
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Presence of chronic pain | Reported at baseline, 3 and 6 months post-injury
  Assessed using a 11-point numerical rating scale from 0 (no pain) - 10 (worst possible pain).
Severity of chronic pain | Reported at baseline, 3 and 6 months post-injury
  Assessed using a 11-point numerical rating scale from 0 (no pain) - 10 (worst possible pain).
Pain impact | Reported at baseline, 3 and 6 months post-injury
  Assessed using the six-item pain interference index

CONTACTS AND LOCATIONS:
Overall Officials: Denise Kendrick, Professor, Study Director — Faculty of Medicine & Health Sciences University of Nottingham; Adam Brooks, FRCS (Gen Surg), Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Queens Medical Centre- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided